CLINICAL TRIAL: NCT03443206
Title: Loves Company: Combatting Emotional Disturbance in the Digital Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: American Psychological Foundation (Other)
Responsible Party: Principal Investigator, Anna Van Meter, Assistant Investigator, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 18-0062-ZHH
Record Dates: First submitted 2018-02-02; First posted 2018-02-23 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Adolescent - Emotional Problem
Keywords: adolescent; mental health; social media
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This condition will include access to a website that includes a social component, in addition to psychoeducation and access to resources.
  Interventions: Other: anonymous social support; Other: psychoeducation; Other: online resources
- Control (Active Comparator): This condition will include access to a website that includes psychoeducation and access to resources.
  Interventions: Other: psychoeducation; Other: online resources

INTERVENTIONS:
Other: anonymous social support — Participants randomized to the intervention condition will be able to communicate with one another and offer social media-based forms of support (e.g., post music, photos, etc).
  Arms: Intervention
Other: psychoeducation — educational materials related to mental health
Other: online resources — links to online mental health resources

SUMMARY:
The goal of this study is to determine whether a community-based website that is intended to provide support for adolescents experiencing psychological distress can improve members' mental health outcomes. The investigators want to understand if a digital platform can help young people who are suffering and may be unlikely to access more traditional forms of mental health services.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-17
* Access to internet-connected device
* Residing in the United States

Exclusion Criteria:

*Inability to assent due to intellectual disability or lack of English language skills

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 212 (Actual)
Dates: Start 2020-06-20 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Adolescent Suicidal Ideation Measure score | 6 months
  frequency of suicidal thoughts and behaviors
Perceived burdensomeness and hopelessness scale score | 6 months
  lower burdensomeness and hopelessness in treatment group (lower score better)
General Behavior Inventory 10D (GBI 10D) | 6 months
  symptoms of depression lower in treatment group (lower score)
Life Satisfaction | 6 months
  level of satisfaction with quality of life

SECONDARY OUTCOMES:
Adolescent Suicidal Ideation Measure score | 12 months
  frequency of suicidal thoughts and behaviors
Perceived burdensomeness and hopelessness scale score | 12 months
  lower burdensomeness and hopelessness in treatment group (lower score better)
General Behavior Inventory 10D (GBI 10D) | 12 months
  symptoms of depression lower in treatment group (lower score)
Life Satisfaction | 12 months
  level of satisfaction with quality of life

OTHER OUTCOMES:
site engagement | 6 months
  time spent on site
General Behavior Inventory 10D (GBI 10D) | weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26
  changes in depressive symptoms
Perceived burdensomeness and hopelessness scale score | weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26
  change in burdensomeness and hopelessness

CONTACTS AND LOCATIONS:
Locations (1):
- Northwell Health, Glen Oaks, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Barzilay S, Feldman D, Snir A, Apter A, Carli V, Hoven CW, Wasserman C, Sarchiapone M, Wasserman D. The interpersonal theory of suicide and adolescent suicidal behavior. J Affect Disord. 2015 Sep 1;183:68-74. doi: 10.1016/j.jad.2015.04.047. Epub 2015 May 7. PMID 26001665
- [Result] Bearman PS, Moody J. Suicide and friendships among American adolescents. Am J Public Health. 2004 Jan;94(1):89-95. doi: 10.2105/ajph.94.1.89. PMID 14713704
- [Result] Belfer ML. Child and adolescent mental disorders: the magnitude of the problem across the globe. J Child Psychol Psychiatry. 2008 Mar;49(3):226-36. doi: 10.1111/j.1469-7610.2007.01855.x. Epub 2008 Jan 21. PMID 18221350
- [Result] Birnbaum ML, Candan K, Libby I, Pascucci O, Kane J. Impact of online resources and social media on help-seeking behaviour in youth with psychotic symptoms. Early Interv Psychiatry. 2016 Oct;10(5):397-403. doi: 10.1111/eip.12179. Epub 2014 Sep 9. PMID 25200743
- [Result] Brissette I, Scheier MF, Carver CS. The role of optimism in social network development, coping, and psychological adjustment during a life transition. J Pers Soc Psychol. 2002 Jan;82(1):102-11. doi: 10.1037//0022-3514.82.1.102. PMID 11811628
- [Result] Gould MS, Velting D, Kleinman M, Lucas C, Thomas JG, Chung M. Teenagers' attitudes about coping strategies and help-seeking behavior for suicidality. J Am Acad Child Adolesc Psychiatry. 2004 Sep;43(9):1124-33. doi: 10.1097/01.chi.0000132811.06547.31. PMID 15322416
- [Result] Heflinger CA, Hinshaw SP. Stigma in child and adolescent mental health services research: understanding professional and institutional stigmatization of youth with mental health problems and their families. Adm Policy Ment Health. 2010 Mar;37(1-2):61-70. doi: 10.1007/s10488-010-0294-z. PMID 20232133
- [Result] La Greca AM, Harrison HM. Adolescent peer relations, friendships, and romantic relationships: do they predict social anxiety and depression? J Clin Child Adolesc Psychol. 2005 Mar;34(1):49-61. doi: 10.1207/s15374424jccp3401_5. PMID 15677280
- [Result] Maher CA, Lewis LK, Ferrar K, Marshall S, De Bourdeaudhuij I, Vandelanotte C. Are health behavior change interventions that use online social networks effective? A systematic review. J Med Internet Res. 2014 Feb 14;16(2):e40. doi: 10.2196/jmir.2952. PMID 24550083
- [Result] McGorry P, Bates T, Birchwood M. Designing youth mental health services for the 21st century: examples from Australia, Ireland and the UK. Br J Psychiatry Suppl. 2013 Jan;54:s30-5. doi: 10.1192/bjp.bp.112.119214. PMID 23288499
- [Result] Safer DJ. Self-reported suicide attempts by adolescents. Ann Clin Psychiatry. 1997 Dec;9(4):263-9. doi: 10.1023/a:1022364629060. PMID 9511952